CLINICAL TRIAL: NCT04472689
Title: Effects of Lidocaine Infusion on Quality of Recovery and Agitation After Functional Endoscopic Sinus Surgery: Randomized Controlled Study
Brief Title: Effects of Lidocaine Infusion on Quality of Recovery and Agitation After Functional Endoscopic Sinus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, rehab zayed, Assisstant Professor of Anesthesia, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0304701
Record Dates: First submitted 2020-07-11; First posted 2020-07-15 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Chronic Polypous Rhinosinusitis
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Active Comparator): patients will receive a loading dose of IV lidocaine 1.5mg/kg slowly diluted with 20 ml normal saline just before induction of anesthesia, then the lidocaine infusion started at a rate of 2mg/kg/h diluted in normal saline by rate of 2 ml/ kg/h.
  Interventions: Drug: Lidocaine
- Control group (Placebo Comparator): patients will receive an equal volume of normal saline (both the loading, and the infusion). The infusion in both groups will be started just after induction of anesthesia induction, and continued until the end of the operation.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — patients will receive a loading dose of IV lidocaine 1.5mg/kg slowly diluted with 20 ml normal saline just before induction of anesthesia, then the lidocaine infusion started at a rate of 2mg/kg/h diluted in normal saline by rate of 2 ml/ kg/h.
  Arms: Lidocaine group
Drug: Normal saline — patients will receive an equal volume of normal saline (both the loading, and the infusion). The infusion in both groups will be started just after induction of anesthesia induction, and continued until the end of the operation
  Arms: Control group

SUMMARY:
The essential anesthesia requirements for FESS include airway management, considerations for facilitating surgical access, provision of a clear and still surgical field for precision surgery, assuring quick and non-stimulating emergence from anesthesia, and fast-tracking patients for discharge. Postoperative agitation, although short-lived, is potentially harmful to both patients and recovery room staff, it has a potential for self-injury by removing intravenous catheters, tubing, oxygen masks and nasal packs. Furthermore, very agitated patients can pose an immediate danger to operating theatre staff.

DETAILED DESCRIPTION:
Lidocaine is an amino amide-type short-acting local anesthetic (LA). It has a short half-life, and a favorable safety profile, and is therefore the LA of choice for continuous IV administration, it has analgesic, and anti-inflammatory effects that are induced by reduction of cytokines production through inhibition of neutrophil activation, and the analgesia may persist even after plasma concentration reduction. It can blunt the pressor response to endotracheal intubation also systemic lidocaine was effective in producing controlled hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective functional endoscopic sinus surgery;
* ASA class I-II,
* aged (20-60 years).

Exclusion Criteria:

* Body mass index >35 kg/m2
* History of allergic reaction to local anesthetic agents especially lignocaine.
* History of preoperative use of opioids.
* Patients with history of uncontrolled hypertension, A-V conduction block.
* History of sleep apnea.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
quality of postoperative recovery | 48hours
  assessed using the Quality of Recovery-40 questionnaire.8, which assesses ﬁve dimensions of recovery
Emergence agitation | 30 minutes postoperative
  using the Richmond agitation-sedation scale

CONTACTS AND LOCATIONS:
Overall Officials: Rehab A. Abd Elaziz, Ass.Prof., Principal Investigator — Alexandria University
Locations (1):
- Rehab Abd Elraof Abd Elaziz, Alexandria, Egypt